CLINICAL TRIAL: NCT06014437
Title: Study on Regeneration of Skin Defects in Diabetic Ulcers Treated With New Electrospun Material Poly (L-lactide-co-caprolactone) and Formulated Porcine Fibrinogen
Brief Title: Study on Regeneration of Skin Defects in Diabetic Ulcers Treated With New Electrospun Material PLCL/Fg
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guili Wang (Other)
Responsible Party: Sponsor-Investigator, Guili Wang, Jinshan hospital Fudan University. Guili Wang is Principal Investigator of vascular surgery, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Jinshan hospital
Record Dates: First submitted 2023-08-17; First posted 2023-08-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Diabetic Foot
MeSH Terms: conditions — Diabetic Foot | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PLCL/Fg (Experimental): Routine ulcerated wounds were cleaned, and the test group was given an equal-sized PLCL/Fg dressing to cover the wounds.
  Interventions: Drug: PLCL/Fg group
- control group (Active Comparator): Routine ulcerated wounds were cleaned and changed, and the control group was given an alginate dressing of equal size to cover the wounds.
  Interventions: Drug: control group

INTERVENTIONS:
Drug: PLCL/Fg group — Routine ulcerated wounds were cleaned, and the test group was given an equal-sized PLCL/Fg dressing to cover the wounds.
  Other Names: PLCL/Fg dressing
  Arms: PLCL/Fg
Drug: control group — Routine ulcerated wounds were cleaned and changed, and the control group was given an alginate dressing of equal size to cover the wounds
  Other Names: alginate dressing
  Arms: control group

SUMMARY:
Prospective cohort studies through clinical trials. Obtained a large amount of real-world data to explore the efficacy of PLCL/Fg dressings for specific clinical applications.

Published 1 relevant SCIE paper. Provide a large amount of data support for the application of PLCL/Fg dressing in diabetic foot ulcer wound repair through basic experimental and clinical experimental studies. It can provide a practical and effective biomaterial for the treatment of clinical skin wound structure and function reconstruction, make the patient's wound healing as soon as possible, benefit the general public, reduce medical expenditure, reduce the burden on the society, lay the foundation for the industrialization and marketization of national innovative medical devices, and help to improve the international status and value of the application.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 90 years; type 1 or type 2 diabetes mellitus; history of ulceration for more than 4 weeks at enrollment; wound area between 1 and 25 square centimeters; wound depth of Wagner grades 1 and 2; and an ABI of 0.7 to 1.3 on the affected lower extremity or a transcutaneous oxygen pressure of greater than or equal to 30 mmHg.

Exclusion Criteria:

* Wound healing percentage greater than 30% during wound preparation (7 days); any infection, osteomyelitis, or other condition that may affect wound healing, such as deep vein thrombosis, rheumatoid arthritis, systemic lupus erythematosus, or any other systemic inflammatory disease.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of complete wound closure during treatment and follow-up (12 weeks). (Outpatient follow-up 2-3 times per week, standardized photographs and measurement of wound size) | 12 weeks
  Complete healing is defined as complete re-epithelialization of the ulcer bed with no discharge. Speed of healing is calculated by measuring the size or percentage reduction in wound area per week.

CONTACTS AND LOCATIONS:
Overall Officials: zhihui dong, Study Chair — Department of Vascular Surgery, Jinshan Hospital, Fudan University
Locations (1):
- Department of Vascular Surgery, Jinshan Hospital, Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
Data will be made available on request.

REFERENCES:
- [Derived] Wang G, Li X, Ju S, Li Y, Li W, He H, Cai Y, Dong Z, Fu W. Effect of electrospun poly (L-lactide-co-caprolactone) and formulated porcine fibrinogen for diabetic foot ulcers. Eur J Pharm Sci. 2024 Jul 1;198:106800. doi: 10.1016/j.ejps.2024.106800. Epub 2024 May 14. PMID 38754593